CLINICAL TRIAL: NCT01944787
Title: Intrapartum Hydration and Rate of Cesarean Delivery Among Nulliparous at > 37 Weeks: A Multicenter Randomized
Brief Title: Hydration and Rate of Cesarean Delivery Among Nulliparous
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chauhan, Suneet P., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-05-SP-50
Record Dates: First submitted 2013-09-06; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine (Active Comparator): IV Hydration at 125 cc hour
  Interventions: Other: Routine
- Intervention (Experimental): IV Hydration at 250 cc hour
  Interventions: Other: IV Hydration at 250cc hour

INTERVENTIONS:
Other: Routine — IV Hydration at 125 cc hour
  Arms: Routine
Other: IV Hydration at 250cc hour — IV Hydration at 250 cc hour
  Arms: Intervention

SUMMARY:
The hypothesis of the present study is the hydration of nulliparous women with 250ml/hour vs. 125ml/hrs would decrease the rate of primary cesarean section.

DETAILED DESCRIPTION:
For this non-blinded randomized clinical trial (RCT) we will recruit approximately 670 women which meet the inclusion criteria across three sites (Eastern Virginia Medical School (EVMS), University of Arkansas for Medical Sciences (UAMS) and Obstetrix Medical Group, in California). When the patient is being scheduled for induction by her physician or when she presents to L&D for induction or in labor, but her cervical dilation on admission is less than 4 cm, the participants will be consented, and then randomized into a study intervention group. Both groups will receive maintenance IV hydration with Lactated Ringer's (LR) solution: Group I will receive LR at 125 ml/hr and group II will receive LR at 250ml/hr. Other than the rate of maintenance IV infusion, the two groups will receive routine intrapartum care.

ELIGIBILITY:
Inclusion Criteria:• Non-anomalous singleton

* Nulliparous (no prior delivery after 20 weeks)
* Presenting at ≥37 weeks of gestation
* Presenting for anticipated induction of labor or spontaneous labor (regular contractions for more than 2 hours), but cervical dilation less than 4 cm
* Rupture of membranes
* Expected to deliver at one of the participating hospitals

Exclusion Criteria:• Not in the inclusion criteria

* Autoimmune disorders (antiphospholipid antibody, lupus, rheumatoid arthritis, scleroderma)
* Diabetes mellitus-gestational or pre-gestational
* Enrollment in another randomized clinical trial
* Hematologic disorders (coagulation defects, sickle cell disease, thrombocytopenia, thrombophilia)
* Hypertension (chronic or pregnancy induced) before randomization
* HIV (human immunodeficiency virus)
* Placenta previa / 3rd trimester bleeding
* Renal insufficiency (serum creatinine > 1.5 mg/dL)
* Restrictive lung disease
* Seizure disorder on medication
* Thyroid disease on medication
* Any contraindications to vaginal delivery (breech, active herpes, schedule cesarean, abnormal fetal heart tracing)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 670 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
rate of cesarean section | 5 Years
  The primary objective of this multi-center RCT is to determine if hydration with 250 ml/hr, when compared to traditional 125 ml/hr, significantly decreases the rate of primary cesarean delivery nulliparous.

SECONDARY OUTCOMES:
labor | 5 Years
  The secondary objectives of this randomized trial are to compare the 2 groups regarding:
  Time from randomization to delivery (minutes)

OTHER OUTCOMES:
The rate of tachysystole (uterine contractions more than 5 in 10 minutes, n/%) | 5 Years
The rate of non-reassuring fetal-heart reassuring tracing treated with terbutaline or other tocolytic agent (n/%) | 5 Years
The indication for cesarean delivery (n/%) versus The indication for operative vaginal delivery (n/%) | 5 Years
Maternal complications (as diagnosed by managing clinician, (n/%) for all): | 5 years
  1. chorioamnionitis
  2. endometritis
  3. wound infection
  4. wound disruption
  5. blood transfusion
Neonatal outcomes (as diagnosed by managing clinician, (n/%) for all): | 5 Years
  1. Apgar score at 1 and 5 min
  2. Birth weight (grams)
  3. Gender (male/female/unknown)
  4. Umbilical arterial pH if available (pH units)
  5. Umbilical arterial base excess if available (mmol/L)
  6. Admission to neonatal intensive care unit (n/%)
  7. Indication for NICU admission (n/%)
  8. Duration of hospitalization (days)
  9. Morbidity defined as one or more of the following as diagnosed by managing physician: Respiratory Distress Syndrome (RDS), Intraventricular Hemorrhage (IVH) grade III/ IV, Necrotizing Enterocolitis (NEC), proven sepsis,seizures (n/%)
  10. Mortality (n/%)
Time of Randomization to complete dilation/ minutes | 5 Years
Time from complete cervical dilation to delivery of newborn/ minutes | 5 years
Time from delivery of newborn to delivery of placenta/ minutes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Suneet P Chauhan, MD, Principal Investigator; Andrew Combs, MD PhD, Principal Investigator — Obstetrix Medical Group
Locations (1):
- C A Combs MD PhD, Campbell, California, United States